CLINICAL TRIAL: NCT03395392
Title: A Randomized, Double-Blind Controlled Comparison of NRX-101 to Lurasidone for Adults With Bipolar Depression and Subacute Suicidal Ideation or Behavior
Brief Title: NRX-101 for Bipolar Depression With Subacute Suicidal Ideation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NeuroRx, Inc. (Industry)
Collaborators: Prevail Infoworks (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX101_003
Expanded Access: NCT05779267 (Available)
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-03

CONDITIONS: Bipolar Depression; Suicidal Ideation and Behavior
Keywords: Bipolar; Cyloserine; Lurasidone; MADRS; CGI-SS; C-SSRS
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation; Behavior | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and Care Providers will be masked with regard to medication administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NRX-101 (Experimental): Following study enrollment and randomization, subjects will receive twice daily NRX-101
  Interventions: Drug: NRX-101
- Lurasidone (Active Comparator): Following study enrollment, subjects will receive twice daily lurasidone
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: NRX-101 — NRX-101, a fixed dose combination of D-cycloserine+lurasidone will be given twice a day by mouth
  Arms: NRX-101
Drug: Lurasidone HCl — Lurasidone HCl will be given twice a day by mouth
  Other Names: Latuda
  Arms: Lurasidone

SUMMARY:
NMDA antagonist drugs have shown to reduce symptoms of depression and suicidal ideation. NeuroRx has developed NRX-101 (fixed dose combination of D-cycloserine and lurasidone) for oral use in the treatment of bipolar depression with suicidal ideation. This study will test the hypothesis that NRX-101 is superior to lurasidone alone (standard of care) in maintaining remission from symptoms of depression (primary endpoint) and suicidal ideation or behavior (declared secondary endpoint) over a six week period of twice-daily oral dosing.

DETAILED DESCRIPTION:
Background and Rationale: NMDA antagonist drugs have shown to reduce symptoms of depression and suicidal ideation. NRX-101 is composed of D-cycloserine (DCS) an NMDA antagonist and lurasidone (5HT2a atypical antipsychotic and antidepressant). In a phase 2 clinical study of bipolar depression and acute suicidal ideation and behavior, (in patients requiring hospitalization) patients received an initial infusion of ketamine and then NRX-101 for 6 weeks. In that phase 2 study, NRX-101 showed the ability to maintain remission from depression and suicidality over 6 weeks when taken twice daily. In this current out patient study, patients with bipolar depression and subacute suicidality (not requiring hospitalization), ketamine will not be used.

Primary Objective:

* To test the hypothesis that treatment with NRX-101 is superior to standard of care (lurasidone) in improving symptoms of depression as measured by the total Montgomery Åsberg Depression Rating Scale (MADRS-10) score in patients with bipolar depression and subacute suicidal ideation and behavior (SSIB) which does not require hospitalization.

Secondary Objectives:

• To test the hypothesis that treatment with NRX-101 is superior to standard of care (lurasidone) in reducing suicidality in depressed bipolar patients with SSIB, as measured by the Columbia Suicide Severity Rating Scale (C-SSRS)

Methodology: : A multi-center, randomized, double-blind, trial in which patients with bipolar depression (MADRS ≥30) and subacute levels of suicidal ideation (C-SSRS 3 or 4, not requiring hospitalization) are randomized to receive twice daily oral NRX-101 or lurasidone (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bipolar disorder by a qualified rater according to the criteria defined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and supported by the Mini International Neuropsychiatric Interview (MINI) 7.0.2.
* Confirmed active suicidal ideation (without the intention to act) as evidenced by an answer of 'Yes' on item 3 and/or item 4 and not requiring hospitalization at Screening and an answer of "No" on item 5 of the C-SSRS.
* A total score greater than or equal to 30 on the 10 items of the MADRS.
* Subject has no co-morbidities as ascertained by medical history, physical examination (including measurement of vital signs), clinical laboratory evaluations, and electrocardiogram (ECG)

Exclusion Criteria:

* Subject has current DSM-5 diagnosis of moderate or severe substance use disorder (except marijuana or tobacco use disorder) within the 12 months prior to Screening.
* Subject has a lifetime history of:

  * phencyclidine (PCP)/ketamine drug abuse, or
  * failed use of ketamine for depression or suicidality.
* Subject has schizophrenia or schizoaffective disorder, or any history of psychotic symptoms when not in an acute bipolar mood episode.
* Subject has a current major psychiatric disorder, diagnosed at Screening
* Subject has been prescribed more than one agent in each of the following categories at randomization:

  * Approved SSRIs
  * Approved serotonin and norepinephrine reuptake inhibitors (SNRIs)
  * Approved tetracyclic antidepressants (TeCAs)
  * Approved Mood stabilizers (e.g., lithium, valproic acid, and lamotrigine)
* Subject has signs and symptoms of active or residual COVID-19, or unresolved symptoms of COVID-19 that impact health

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in MADRS-10 over 42 Days | Six weeks
  Mean change from baseline to endpoint (Day 42/exit) in total MADRS score, a 10-item clinician-rated scale, with each item rated on a 0-6 severity scale (0 Minimum, 60 maximum), where higher scores indicate a worse outcome

SECONDARY OUTCOMES:
Mean Change from baseline in CGI-SS | Six Weeks
  Mean change from baseline to exit (Day 42/exit) in CGI-SS score
Time to Treatment Failure | 6 weeks
  Time to relapse, where relapse is defined as experiencing a return of suicidality in the Columbia Suicide Severity Rating Scale (C-SSRS) of >=4)), or a return to baseline levels of depression following an improvement of 25% or greater on the MADRS score, or the need to implement a new treatment plan. The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed in the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. A lower score on the C-SSRS indicates a better outcome (min=0, max=5)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brecher, MD, Study Director — NRx Pharma; Andrew A Nierenberg, MD, Study Chair — Harvard Medical School (HMS and HSDM); Jonathan C Javitt, MD, MPH, Study Chair — NRx Pharmaceuticals
Locations (14):
- United States (14):
  - Science 37, Culver City, California
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - ACMR, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - iResearch Savannah, Savannah, Georgia
  - CBH Health, Gaithersburg, Maryland
  - Omaha Insomnia and Psychiatric Services, Omaha, Nebraska
  - Dent Neurologic Institute, Amherst, New York
  - Peace Health Medical Group, Eugene, Oregon
  - University of Texas Health Austin, Austin, Texas
  - Roots Behavioral Health, Austin, Texas
  - JPS Health, Fort Worth, Texas
  - Houston Mind and Brain, Houston, Texas
  - Health Texas, Richmond, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared under an approved confidentiality agreement within one year of drug approval
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year of drug approval
URL: http://nrxpharma.com

REFERENCES:
- [Derived] Sapko MT, Kolesar C, Sharp IR, Javitt JC. Quality Assurance of Depression Ratings in Psychiatric Clinical Trials. J Clin Psychopharmacol. 2025 Jan-Feb 01;45(1):28-31. doi: 10.1097/JCP.0000000000001936. Epub 2024 Nov 21. PMID 39714786
- See also: STABIL-B Study Results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10423711/
- See also: Data Quality Assessment — https://papers.ssrn.com/sol3/papers.cfm?abstract_id=4537055

DOCUMENTS (2):
  • Study Protocol (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03395392/Prot_001.pdf
  • Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03395392/SAP_002.pdf